CLINICAL TRIAL: NCT06621823
Title: Image-guided Ultrasound Robotic Intraoperative Evaluation of Lymph-nodes Status in Gynecological Malignancies
Acronym: R-LYNUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6534
Record Dates: First submitted 2024-05-20; First posted 2024-10-01 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Lymph Node Metastasis; Gynecologic Cancer
MeSH Terms: conditions — Lymphatic Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- surgical lymph nodes (Other): Patients referred to the Gynecology Oncology Unit in Fondazione Policlinico A. Gemelli IRCCS, Italy, Rome with a diagnosis of gynecological malignancy requiring surgical lymph nodes harvest will be evaluated for the enrolment.
  Interventions: Procedure: image-guided surgery technique

INTERVENTIONS:
Procedure: image-guided surgery technique — The identification of an image-guided surgery technique capable of intraoperatively detecting the presence of lymph node metastases would overcome the disadvantages and complications of extensive staging lymphadenectomies.

SUMMARY:
The assessment of lymph node status is of crucial importance in gynaecological malignancies.

Indeed, the prognosis and adjuvant treatment regimens are strongly influenced by the presence of nodal involvement. Systematic extensive lymphadenectomies are often performed for staging, diagnosis of skip metastases and to define the radiation field when radiotherapy treatments are required. Nevertheless, these can lead to significant short-term and long-term lymphatic complications, which are difficult to justify if the lymph nodes are free from metastasis. To avoid unnecessary comprehensive procedures in early-stage cancers, evaluation of the sentinel lymph node has acquired a valuable role even if limitations are still present (rate of frozen section false negative, "empty packets" and mapping failure). The introduction of an intra-operative non-invasive imaging technique capable of describing the presence and characteristics of lymph nodes could help in (1) eliminating the risk of empty packet, (2) orienting the intraoperative decision while avoiding the drawbacks of frozen section (time and resources, partial destruction of the tissue material), (3) orientate the pathological section if frozen section is used. To date, technological advancements have paved the way for enhanced intra-operative assessment of cancerous organs and lesions. Over the past decade, the evolution of robotic surgery combined with advancements in image-guided surgery techniques has led to the introduction of ultrasound probes designed specifically for intraoperative ultrasound during robotic surgery (RIOUS). Apart from the conventional rigid laparoscopic probes, which can be inserted through an accessory trocar, there are robotic probes tailored to fit device arms, and drop-in flexible probes that are becoming increasingly relevant in the scientific panorama. Notably, the latter drop-in probes feature a rigid segment designed for compatibility with robotic graspers, leveraging the dexterity and rotational manoeuvrability inherent to robotic surgery. Such probes, already proven effective in evaluating liver and kidney lesions as well as tumour margins, hold promise for intraoperative lymph node assessments due to the possibility of reaching difficult anatomical spaces thanks to the robotic-assisted movements

DETAILED DESCRIPTION:
Women undergoing radical surgery for gynecological cancers who meet the inclusion criteria in absence of exclusion criteria will be considered candidate for the study. Intraoperative robotic ultrasound will be performed on in vivo lymph nodal samples. Lymph nodes morphology and imaging characteristics will be evaluated. The gold standard will be definitive pathology.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing robotic surgery for gynecological malignancies (ovarian, endometrial, cervical cencers)
* Need for nodal excision (staging or cytoreductive reasons)
* 18-99 years old
* Absence of contemporary lymphatic diseases
* Absence of previous oncological disease in the last 5 years
* Willingness to participate in the study and to provide informed consent

Exclusion Criteria:

* - Previous radiotherapy treatments in the area of analysed lymph nodes
* Previous chemotherapy treatments

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of RIUS in detecting lymph node metastases (macro-, micro-metastases and isolated tumor cells) | 2 year
  The aim of this prospective trial is to evaluate the sensitivity of Real-time Intraoperative Ultrasound (RIUS) in detecting lymph node metastases, including macrometastases, micrometastases, and isolated tumor cells (ITCs), using fresh, unstained in vivo lymph node samples. Ultrasound images will be assessed according to the VITA (Vulva International Tumor Analysis) group consensus on morphological parameters. Final histopathological examination will serve as the gold standard for comparison.

SECONDARY OUTCOMES:
drop-in robotic ultrasound probe | 2 years
  The secondary endpoint is to assess the lowest size detectable with the adopted drop-in robotic ultrasound probe

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Carla Testa, Professor, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome; Francesco Fanfani, Professor, Study Chair — Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome; Matteo Pavone, MD, Study Chair — Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome; Elena Teodorico, MD, Study Chair — Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome; Denis Querleu, Professor, Study Chair — Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome; Giovanni Scambia, Professor, Study Director — Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

REFERENCES:
- [Derived] Pavone M, Teodorico E, Bizzarri N, Innocenzi C, Rosati A, Zorzi M, Cantarini C, Ciancia M, Moro F, Gallotta V, Marescaux J, Lecointre L, Fagotti A, Scambia G, Fanfani F, Testa A, Querleu D. Image-Guided Robotic Surgery for Sentinel Lymph Node Status Assessment in Uterine Cancers Using Ultrasound Drop-in Probe: Surgical Technique in 10 Steps. Ann Surg Oncol. 2025 May;32(5):3465-3466. doi: 10.1245/s10434-025-16912-x. Epub 2025 Feb 1. PMID 39893338

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT06621823/Prot_SAP_000.pdf